CLINICAL TRIAL: NCT00431054
Title: Pharmacodynamic Trial: Molecular Marker & Imaging Studies as Primary Endpoints to Determine Optimal Biological Dosage of Perifosine, Orally Avail AKT PH Domain Inhibitor Combined w/ Docetaxel in Patients w/Relapsed Epithelial Ovarian Cancer
Brief Title: Perifosine and Docetaxel in Patients With Relapsed Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0970
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2012-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Perifosine; Docetaxel; Taxotere
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — perifosine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perifosine + Docetaxel (Experimental)
  Interventions: Drug: Perifosine; Drug: Docetaxel

INTERVENTIONS:
Drug: Perifosine — Loading Dose = 100 mg by mouth (PO) every 6 hours, followed by 50 mg by mouth (PO) daily
Drug: Docetaxel — 75 mg/m^2 by vein over 1 hour every 4 weeks
  Other Names: Taxotere

SUMMARY:
The goal of this clinical research study is to find out if a combination treatment of perifosine and docetaxel will help shrink or slow the growth of cancer cells in recurrent ovarian cancer. The safety of this combination treatment will also be studied.

DETAILED DESCRIPTION:
Docetaxel is a chemotherapy drug designed to kill some cancers and is believed to be slightly effective at killing blood vessels in cancers.

Perifosine is a new drug that may help docetaxel be more effective in causing cancer cells to die. Perifosine alone may slow cancer cell growth by targeting an abnormal pathway in your ovarian cancer cells.

If you are found to be eligible to take part in this study, you will receive your dose of perifosine by mouth every 6 hours on Day 1 of therapy. The actual number of pills in your dose depends upon which dose level you are assigned to. You will then continue receiving perifosine by mouth once a day for 20 more days. Each cycle of treatment is about 28 days.

On Day 5 of therapy, of the first cycle only, you will have blood drawn (about 2.5 tablespoons) performed, and 5 hair follicles and ascites collected, if available. If you do not have ascites, you will have a FNA performed on your tumor.

On Day 8 of therapy, you will have a DCE-MRI. On Day 10 of therapy, you will have a PET scan. Your treatment schedule for each cycle will usually be the same. There may be a one-day difference in the treatment schedules.

After the first cycle is completed, you will begin receiving docetaxel, on Day 2 of therapy of each cycle of treatment, as an injection in a vein over 60 minutes at the M. D. Anderson infusion center. The second cycle of treatment will start on Day 29.

Within 72 hours of the start of each cycle, you will have blood (about 1 tablespoon) and urine collected for routine tests . After you receive the drugs, you will have weekly blood tests (about 1 tablespoon) to evaluate your well being. Before the start of each cycle of therapy, you will have a physical exam, and your medical history will be recorded. You will also be called by the study doctor or staff to ask questions about any side effects you may be experiencing during therapy. After the end of every 2 cycles (about every 8 weeks), you will have an x-ray and either a CT scan or an MRI to re-evaluate your cancer.

You may be given treatment on this study as long as your disease does not get worse. Your physician will discuss with you the maximum number of treatment cycles you will receive. You will be taken off this study if your disease gets worse or if you experience any intolerable side effects.

After your participation in this study has ended, you will come back for a follow-up visit. At this visit, you will have your medical history recorded and a physical exam. You will have blood (about 1 tablespoon) and urine collected for routine tests. You may also have a CT scan or an MRI to re-measure and re-evaluate your cancer.

You will have follow-up for as long as needed after you have completed treatment with perifosine plus docetaxel. You will either be contacted by phone or asked to come to the clinic for a routine visit. You will be contacted every 8 weeks. You will have radiographic evaluations, by either a CT or an MRI, done every 12 weeks to evaluate your cancer growth or until you start on another anticancer therapy.

This is an investigational study. Perifosine has been authorized by the FDA for use in research only. Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically or cytologically confirmed diagnosis of epithelial cancer of the ovary, fallopian tube cancer or gynecologic primary peritoneal cancer. All patients must be platinum resistant or refractory that is defined as tumor progression during platinum-based treatment or less than 6 months of treatment-free interval.
2. All patients have to have tumor that is accessible to biopsy. In addition, patients have to have another tumor that a) will not be biopsied; and for the purpose of DCE-MRI and PET studies, b) is at least 2cm in size per radiologic measurement.
3. Patient is at least 18 years of age.
4. Patient has an ECOG performance status of 0-2.
5. Patient is willing to comply with study procedures to have biopsies of tumor and blood collection for molecular marker and biological marker studies; and two PET scans and two dynamic MRIs for imaging studies and follow-up examinations for toxicity profile.
6. Patients must be informed of the investigational nature of this study and give written IRB-approved informed consent according to institutional guidelines.
7. If patient is of child-bearing potential, she has agreed to practice an effective method of birth control during the study and 6 months after the last study dose.
8. Patient has adequate liver and renal function: serum bilirubin =/<2.0 mg/dL; ALT=/<3x uln. If the patient has hepatic metastasis, ALT =/<5x uln. Serum creatinine =/<2.0 mg/dL or a calculated creatinine clearance of at least 50 ml/min.
9. Patient has adequate bone marrow reserve. ANC=/>1,500/mm^3, Platelet count =/>100,000/mm^3, and Hemoglobin =/>9.0g/dL without bone marrow support.

Exclusion Criteria:

1. Any concurrent chemotherapy.
2. Underlying medical condition that might be aggravated by treatment or that cannot be controlled, i.e. active uncontrolled infection and cardiac dysfunction.
3. Medical and psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk.
4. Known hypersensitivity to study drugs or its analogs.
5. Failure to recover from any prior surgery within 4 weeks of study entry.
6. Pregnant or lactating.
7. On combination anti-retroviral therapy for HIV because of possible pharmacokinetic interaction with perifosine. Every effort will be made to avoid known inhibitors or inducers of P450 enzymes for potential drug-drug interaction.
8. Any treatment specific for tumor control within 3 weeks of study drugs (within 6 wks. for nitrosoureas or mitomycin C) or failure to recover from the toxic effect of any of these therapies prior to study entry.
9. Any signs of intestinal obstruction interfering with nutrition. Patient cannot tolerate oral intake for any reason.
10. A known history of CNS metastasis unless the patient has had treatment with surgery or radiation therapy, is neurologically stable, and does not require oral or intravenous corticosteroids or anticonvulsants.
11. Any investigational drug within 30 days of first day of dosing.
12. History of high-dose chemotherapy for ovarian cancer, defined as the intensity and/or the density of a chemotherapeutic agent beyond standard of care for ovarian cancer treatment. i.e. Treatment with carboplatin at AUC 11 is considered as high-dose chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Tumor Response | After the end of every 2 cycles (about every 8 weeks), an x-ray and either a CT scan or an MRI will be obtained to re-evaluate tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org